CLINICAL TRIAL: NCT04074564
Title: An Exploratory Study Evaluating the Safety and Efficacy of MASCT-I Combined With Apatinib Mesylate and/or Camrelizumab in the Treatment of Patients With Advanced Bone and Soft Tissue Sarcoma
Brief Title: MASCT-I Combined With Apatinib and/or Camrelizumab in the Treatment of Bone and Soft Tissue Sarcoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HRYZ Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASCT-I-1005
Record Dates: First submitted 2019-08-26; First posted 2019-08-30 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Sarcoma
Keywords: MASCT-I; Cell-based immunotherapy; Camrelizumab; Apatinib; Tumor associated antigen
MeSH Terms: conditions — Sarcoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (Experimental): Subgroup 1: MASCT-I A+Camrelizumab+Apatinib combination therapy; Subgroup 2: MASCT-I B+Camrelizumab+Apatinib combination therapy
  Interventions: Combination Product: MASCT-I, Camrelizumab,Apatinib
- Part B (Experimental): MASCT-I (based on the administration schedule selected from part A) in combination with Apatinib
  Interventions: Combination Product: MASCT-I, Camrelizumab,Apatinib

INTERVENTIONS:
Combination Product: MASCT-I, Camrelizumab,Apatinib — Multi-Antigen Stimulated Cell Therapy-I Injection (MASCT-I) is a sequential immune cell therapy.
  Camrelizumab is an immune checkpoint inhibitors against PD-1.
  Apatinib is a highly selective tyrosine kinase inhibitor targeting VEGFR2.

SUMMARY:
This study will evaluate the safety and preliminary efficacy of Multi-Antigen Stimulated Cell Therapy-I Injection (MASCT-I) in combination with Apatinib and/or Camrelizumab in patients with advanced bone and soft-tissue sarcoma.

DETAILED DESCRIPTION:
This is a single-center, open-label, exploratory study to evaluate the safety, preliminary efficacy and immune response of MASCT-I with Apatinib and/or Camrelizumab in the treatment of patients with advanced bone and soft-tissue sarcoma. 60 patients with advanced bone and soft-tissue sarcoma will be recruited.

This study include two parts. In part A, patients were randomized into two groups: one group received MASCT-I A+Camrelizumab+Apatinib, and the other group received MASCT-I B +Camrelizumab+Apatinib, the administration schedules for MASCT-I is different between two groups. A total of 20 patients were planned to be recruited in part A. In part B, patients will be treated with MASCT-I (based on the administration schedule selected from part A) in combination with Apatinib. 40 patients were planned to be recruited in part B.

MASCT-I A and MASCT-I B were administered mainly at different frequencies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 14-70 years old.
2. Obtain the written informed consent of the patient/legal representative;
3. In patients with unresectable recurrent or metastatic advanced bone and soft tissue sarcoma, histologically or cytologically confirmed objective radiographic progression (RECIST 1.1) after first-line or further lines treatment, and the maximum diameter of metastatic lesions is ≤ 8 cm. When objective radiographic progression (RECIST 1.1) found in patients with alveolar soft-part sarcoma and clear cell sarcoma, even if they have not received first line or further lines treatment could also be included in this study;
4. The interval between the last PD-1/PD-L1/CTLA-4 antibody treatment and enrollment was more than 4 weeks;
5. At least one measurable and assessable lesion defined by RECIST 1.1;
6. ECOG performance status of 0-1 (2 for amputees);
7. Estimated life expectancy ≥ 6 months;
8. At least 4 weeks after the last chemotherapy;
9. Cardiopulmonary function is basically normal.
10. Tumor tissue specimens could be provided for PDL1, MSI detection.
11. Blood samples could be provided for immune response test.
12. Patients with potential fertility need to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill or condom) during the study treatment period and within 6 months after the end of the study treatment period; The serum or urine HCG test must be negative within 72 hours before the study was included; And must be non lactating.
13. Patients with organ function as defined below (any blood components and growth factors are not allowed within 14 days before screening):

A) Hemoglobin ≥ 90g/L;

B) Leukocyte ≥3.0 *109/L;

C) The absolute neutrophil count (ANC) ≥ 1.5 x 109/L;

D) Platelet ≥ 70 *109/L;

E) ALT, AST ≤ 2.5 ULN (Upper Limit of Normal);

F) ALP ≤ 2.5 ULN;

G) Serum total bilirubin < 1.5 ULN; Patients with Gilbert's syndromes (persistent or repeated hyperbilirubinemia [mainly unconjugated bilirubin], in the absence of evidence of hemolysis or liver disease), are allowed to consult a doctor.

H) Serum urea nitrogen and creatinine ≤ 1.5 ULN;

I) Serum albumin ≥30g/L.

Exclusion Criteria:

1. Subjects have participated in another clinical study at the same time, observational studies are not included.
2. Those who have received other systemic anti-tumor treatment.
3. Pregnant or plan to get pregnant.
4. Allergic to sodium citrate or human albumin.
5. Those with brain metastases ( Brain metastases confirmed by imaging, inactive, asymptomatic, whether or not treated, and stable for more than 6 months can be included);
6. Subjects have received MASCT or other cellular immunotherapy in the past 1 year.
7. Subjects with severe coagulation dysfunction (PT, TT, APTT or fibrinogen was found to be abnormal and have clinical significance).
8. Subjects have undergone significant bleeding symptoms or bleeding tendency within 3 months before enrollment, or have undergone arterial/venous thrombotic events within 6 months before enrollment. Subjects with long-term anticoagulation of warfarin or heparin or long-term antiplatelet therapy (aspirin ≥300mg/ day or clopidogrel ≥75mg/ day) are not included in this study.
9. Allogeneic organ transplanters, including bone marrow transplantation and peripheral stem-cell transplantation, corneal transplantation is not included.
10. Subjects were using immunosuppressive agents or systemic or absorbable local hormones to achieve immunosuppressive purposes (dose > 10mg/day of prednisone or other therapeutic hormones) and were still using them within 2 weeks before enrollment.
11. Systematic or long-term use of immunomodulators such as interferon, thymosin and immunosuppressive drugs such as adrenocorticosteroids in half a year; Systematic or long-term use of immunomodulators for more than three months and immunosuppressive drugs for more than one month;
12. Subjects have any active autoimmune disease or history of autoimmune disease.
13. Subjects with active tuberculosis.
14. Subjects who have undergone major surgery within 28 days before 1st treatment (according to the investigator's definition);
15. Subjects were infected with hepatitis B virus, hepatitis C virus or HIV, or syphilis.
16. Subjects with or have history of peripheral nervous system disorders or mental disorders.
17. Subjects have active infection or fever of unknown cause during screening and before 1st treatment more than 38.5 degrees (patients with fever caused by cancer is eligible for enrollment according to investigator's judgement);
18. Chronic systemic diseases such as severe liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease, or diabetes mellitus (fasting plasma glucose > 7.0mmol/L or 2-hour postprandial plasma glucose >11.1mmol/L) that cannot be well controlled by medical treatment, hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90mmHg);
19. Subjects with other malignant tumors (except cured skin basal cell carcinoma, thyroid carcinoma and cervical carcinoma in situ) within 5 years before enrollment or at enrollment;
20. Subjects with poorly controlled cardiac symptoms or diseases, such as: (1) heart failure of NYHA class 2 or higher (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention (5) LVEF<50% (6) poorly controlled arrhythmias (QTcF interval > 450ms for men and > 470ms for women);
21. According to investigator's judgement, those who are not suitable for enrollment.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2024-08-07 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events (safety) | 4 years
  All adverse events and serious adverse events during the study

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 4 years
  The percentage of participants with complete response (CR) or partial response (PR) via investigator assessment per RECIST (Response Evaluation Criteria In Solid Tumors Criteria) v1.1 relative to the total number of participants in the analysis population.
Progression-Free Survival (PFS) | 4 years
  The time from the date of randomization to the first occurrence of radiological progression or death, whichever comes first.
Disease Control Rate (DCR) | 4 years
  The percentage of participants with CR, PR, or stable disease (SD) relative to the total number of participants within the analysis population as determined by Investigators per RECIST v1.1.
Overall Survival (OS) | 4 years
  The interval of time between the date of enrollment and the date of death.
immune response | 4 years
  Specific immune responses to tumor-associated antigens were detected at different time points according to different administration schedules.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou Y, Li M, Zhang B, Yang C, Wang Y, Zheng S, Tang L, Zhou C, Qian G, Huang Y, Yu W, Li H, Wang Y, He A, Shen Z, Zhang J, Li X, Yang Q, Hu H, Yao Y. A pilot study of multi-antigen stimulated cell therapy-I plus camrelizumab and apatinib in patients with advanced bone and soft-tissue sarcomas. BMC Med. 2023 Nov 29;21(1):470. doi: 10.1186/s12916-023-03132-x. PMID 38031088